CLINICAL TRIAL: NCT02196922
Title: Telehealth Self-Management Program in Older Adults Living With Heart Failure in Health Disparity Communities
Brief Title: Telehealth Management in HF Disparity Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Renee Pekmezaris, principal investigator, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCT02196922
Record Dates: First submitted 2014-07-18; First posted 2014-07-22 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Chronic Heart Failure
Keywords: Chronic Heart Failure; Telehealth; Self Management
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (Active Comparator): Patients in the control group will receive standard of care at a Heart Failure clinic (primary and cardiac care as reimbursed by Medicare or sliding scale/uncompensated care). Standard of care patients will be contacted on a weekly basis in order to maintain comparable frequency of contact.
  Interventions: Other: Standard of Care
- Telehealth Self Management (TSM) (Experimental): TSM is defined as a weekly clinical telehealth visit and self-monitoring of daily vital signs utilizing a subject monitor which connects from the subject's residence, via a standard telephone line to the provider station.
  Interventions: Device: Telehealth Self Management (TSM)

INTERVENTIONS:
Device: Telehealth Self Management (TSM) — Experimental: Telehealth Self Management (TSM) TSM is defined as a weekly clinical telehealth visit and self-monitoring of daily vital signs utilizing a subject monitor which connects from the subject's residence, via a standard telephone line to the provider station.
  Arms: Telehealth Self Management (TSM)
Other: Standard of Care — Patients receiving standard of care experience typical chronic care management received by Medicare patients.
  Arms: Standard of Care

SUMMARY:
In the US, racial and ethnic disparities persist, even when income, health insurance and care access are addressed. For example, there is a greater prevalence of chronic heart failure (CHF), higher rates of hospital use and higher death rates in blacks as compared to whites. This is due to many factors including: reduced healthcare access, higher prevalence of hypertension,coronary artery disease, systolic dysfunction, myocardial infarction and obesity. Given the magnitude of this chronic health issue, the growth of the elderly population, and increases in ethnic diversity, providers need to develop new ways of caring for those with chronic conditions living in health disparity communities.

The investigators propose to implement a randomized study with health disparity community-dwelling patients. A bilingual clinician will follow patients for 3 months after hospitalization for CHF to test this approach for the proposed health disparity population. The investigators will obtain patient/caregiver input at multiple points during the research to make necessary adjustments to the intervention to ensure that disparity patients accept/use the system, and are satisfied. To ensure that proposed outcomes have relevance for patients, a Community Advisory Board (CAB) of stakeholders will advise the study team throughout the study process. The investigators believe that studying patient use of TSM over a 3 month period will: 1) identify cost-effective care approaches for patients living with chronic disease; 2) involve the patient in identifying and testing approaches that work for them; 3) enhance provider-patient communication; 4) teach the patient how to self-monitor and explore his/her role in self-care; 5) improve patient education about treatment options and 6) explore how "usable" the patients feel the program is. If our goals are achieved, these strategies will result in patient-led improvements in health, satisfaction and quality of life. Knowledge gained will further understanding of the use of telehealth programs as effective self-management tools.

DETAILED DESCRIPTION:
Disparities in cardiovascular disease have received particular focus, as cardiovascular disease is a major contributor to differences in morbidity and mortality between blacks and whites. African Americans, for example, are hospitalized for chronic heart failure (CHF) at a higher rate than whites and are 30% more likely to die from CHF than white individuals. Community-dwelling patients with CHF typically receive exacerbation-focused care, leading to high rates of emergency department (ED) and hospital utilization. The lack of comprehensive chronic disease management leads to poor patient outcomes, and increased health care costs. Given the larger burden of CHF and the unfavorable disease outcomes in disparity communities, a tailored and more focused management of this clinical condition is warranted.

We propose to:

1. Assess telehealth self management (TSM) usability, utilizing a mixed-methods approach, focusing on patient and stakeholder input, with the goal of adapting the intervention to facilitate acceptability and feasibility in a population of low-income ethnic minority patients. Prior to intervention implementation, we will determine characteristics of the intervention requiring adaptation to maximize usability through focus groups, with key community stakeholders, patients and caregivers. We will continue the qualitative usability assessment during the intervention with patients enrolled in the study to identify barriers/challenges to usability, to further adapt the intervention. Finally, we will use quantitative methods to assess usability. These quantitative indicators will also be used to make adjustments and inform future wide-scale interventions that will be conducted in this community.
2. Compare hospital utilization of low income ethnic minority patients receiving telehealth technology vs. demographically matched patients receiving standard of care. A randomized controlled clinical trial will be conducted to test the primary hypothesis that health care utilization will be lower in the in the TSM group than the usual-care group. We will specifically compare acute care and ED utilization and quality of life (Minnesota QoL Questionnaire) between groups. We will adjust for potential confounders (demographic, clinical, educational and functional/support variables). The target population is community-dwelling CHF patients discharged home from the Nassau University Medical Center.

This research will further our understanding of the use of TSM in the management of CHF for low income, ethnic minority seniors. The proposed research will improve patient outcomes while reducing unnecessary hospitalizations and ED burden. Chronic disease self-management programs have the potential to reduce health care costs while improving patient health status, particularly for medically underserved communities.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Heart Failure (CHF) patients about to be discharged from Nassau University Medical Center (NUMC)
* 18 years and older
* New York Heart Association (NYHA) class of 1-3
* Primary language of Spanish or English
* Access to a phone (land line or cell),
* Folstein Mini Mental Status Exam (MMSE) score of 21 or higher.

Exclusion Criteria:

* Patients with heart failure NYHA class 4
* Patients under age 18
* Anyone with a primary language that is not English or Spanish
* Anyone with a Folstein MMSE score under 21 (indicative of cognitive impairment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2014-01-01; Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renee Pekmezaris, PhD, Principal Investigator — Northwell Health
Locations (1):
- Nassau University Medical Center, East Meadow, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pekmezaris R, Schwartz RM, Taylor TN, DiMarzio P, Nouryan CN, Murray L, McKenzie G, Ahern D, Castillo S, Pecinka K, Bauer L, Orona T, Makaryus AN. A qualitative analysis to optimize a telemonitoring intervention for heart failure patients from disparity communities. BMC Med Inform Decis Mak. 2016 Jun 24;16:75. doi: 10.1186/s12911-016-0300-9. PMID 27343060

RESULTS

PARTICIPANT FLOW:
Groups:
- Comprehensive Outpatient Management (COM-Standard of Care): Patients in the control group will receive comprehensive outpatient management (COM)at a Heart Failure clinic (primary and cardiac care as reimbursed by Medicaid, Medicare or sliding scale/uncompensated care). COM patients will be contacted on a weekly basis in order to maintain comparable frequency of contact.
  COM: Patients receiving COM experience chronic care management received by disparity patients at a heart failure clinic.
- Telehealth Self Management (TSM): Telehealth Self Management (TSM): Experimental: TSM is defined as a weekly clinical telehealth visit and self-monitoring of daily vital signs utilizing a subject monitor which connects from the subject's residence to the provider station.
Period: Overall Study
Arm/Group | Comprehensive Outpatient Management (COM-Standard of Care) | Telehealth Self Management (TSM)
Started | 58 | 46
Completed | 58 | 46
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Comprehensive Outpatient Management (COM): Patients in the control group will receive COM at a Heart Failure clinic (primary and cardiac care as reimbursed by Medicaid, Medicare or sliding scale/uncompensated care). COM patients will be contacted on a weekly basis in order to maintain comparable frequency of contact.
  COM: COM experience typical chronic care management received by disparity patients I a heart failure clinic.
- Telehealth Self Management (TSM): Telehealth Self Management (TSM): Experimental is defined as a weekly clinical telehealth visit and self-monitoring of daily vital signs utilizing a subject monitor which connects from the subject's residence to the provider station.
- Total: Total of all reporting groups
Arm/Group | Comprehensive Outpatient Management (COM) | Telehealth Self Management (TSM) | Total
Number analyzed (Participants) | 58 | 46 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (15.0) | 58.4 (15.2) | 59.9 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 20 | 43
  Male | 35 | 26 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 15 | 32
  Not Hispanic or Latino | 41 | 31 | 72
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 41 | 31 | 72
  White | 17 | 15 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 58 | 46 | 104

OUTCOME MEASURES:

1. Primary Outcome: Hospitalizations
Description: Number of hospitalizations during the 90 day observation period
Time Frame: Baseline and Day 90
Population: Intention to treat population (all participants who are randomized to either COM or TSM.
Measure: Mean (Standard Deviation); unit: participant mean hospitalizations/90 day
Groups:
- Comprehensive Outpatient Management (COM): Patients in the COM group will receive outpatient care at a Heart Failure clinic (primary and cardiac care as reimbursed by Medicaid, Medicare or sliding scale/uncompensated care). COM patients will be contacted on a weekly basis in order to maintain comparable frequency of contact.
  COM: Patients receiving COM experience typical chronic care management received by disparity patients at heart failure clinic.
Arm/Group | Comprehensive Outpatient Management (COM) | Telehealth Self Management (TSM)
Number analyzed (Participants) | 58 | 46
participant mean hospitalizations/90 day | .55 (0.9) | .78 (1.3)

2. Primary Outcome: Emergency Department Visits
Description: Emergency Department Visits, defined as Mean Number of visits over the 90 day observation period
Time Frame: Days 0-90
Population: Intention to Treat population (all participants to COM or TSM)
Measure: Mean (Standard Deviation); unit: participants group mean ED visits/90 day
Groups:
- Comprehensive Outpatient Management (COM): Patients in the COM group will receive outpatient management at a Heart Failure clinic (primary and cardiac care as reimbursed by Medicaid, Medicare or sliding scale/uncompensated care). COM patients will be contacted on a weekly basis in order to maintain comparable frequency of contact.
  Patients receiving COM experience typical chronic care management received by disparity patients at a heart failure clinic.
- Telehealth Self Management (TSM): Telehealth Self Management (TSM): Experimental: is defined as a weekly clinical telehealth visit and self-monitoring of daily vital signs utilizing a subject monitor which connects from the subject's residence, to the provider station.
Arm/Group | Comprehensive Outpatient Management (COM) | Telehealth Self Management (TSM)
Number analyzed (Participants) | 58 | 46
participants group mean ED visits/90 day | .69 (.99) | .63 (1.18)

3. Secondary Outcome: Quality of Life
Description: Minnesota Quality of Life Questionnaire is a validated instrument specifically designed to measure quality of life for heart failure patients. Possible scores range from 0 (best quality of life) to 105 (worst quality of life)
Time Frame: Baseline and Day 90
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Comprehensive Outpatient Management (COM) | Telehealth Self Management (TSM)
Number analyzed (Participants) | 58 | 46
units on a scale | 27.8 [0 to 105] | 36.3 [0 to 105]

ADVERSE EVENTS:
Time Frame: days 0-90
Arm/Group | Comprehensive Outpatient Management (COM) | Telehealth Self Management (TSM)
All-Cause Mortality (participants affected / at risk) | 1/58 | 1/46
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/46
Other Adverse Events (participants affected / at risk) | 0/58 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-03-25): https://cdn.clinicaltrials.gov/large-docs/22/NCT02196922/Prot_000.pdf
  • Statistical Analysis Plan (2016-03-25): https://cdn.clinicaltrials.gov/large-docs/22/NCT02196922/SAP_001.pdf